CLINICAL TRIAL: NCT03763435
Title: The Effects of Pregnancy Classes on Postpartum Depression and Contributing Factors to Postpartum Depression
Brief Title: The Effects of Pregnancy Classes and Contributing Factors to Postpartum Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bartin State Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Yassa, Principal Investigator, Bartin State Hospital
Other Study IDs: Bartin2018-3
Record Dates: First submitted 2018-11-24; First posted 2018-12-04 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Postpartum Depression; Sleep Disorder; Breast Feeding; Self Esteem
Keywords: postpartum depression; sleep disorder; genital self-image; breast-feeding; prevalence
MeSH Terms: conditions — Depression, Postpartum; Sleep Wake Disorders; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antenatal Classes Received: Women who are involved into at least 3 comprehensive session of Antenatal pregnancy classes (educational) during the prenatal period.
  Interventions: Behavioral: Antenatal pregnancy classes
- Without education: Groups are not randomized for not to give rise to ethical problems in order to maximize the community health care. Only women who are not involved into the educational classes due to their inaccessibility related to their own conditions or wishes.

INTERVENTIONS:
Behavioral: Antenatal pregnancy classes — At least three comprehensive full-day educational program covering all the stages of pregnancy.
  Groups: Antenatal Classes Received

SUMMARY:
It is recommended by the American College of Obstetricians and Gynecologists' Committee on Obstetric Practice that all obstetricians screen each women for postpartum depression and anxiety with a validated instrument. Although much effort is made, the contributing factors still lack in the literature due to its multi-factorial nature and complexity.

In addition, the effects of prenatal education classes remain understudied. Therefore, this study aims to demonstrate the prevalence, characteristics and contributing factors of the postpartum depression. In addition, the change in prevalence and characteristics of the postpartum depression among women who had prenatal classes and not will also be assessed.

DETAILED DESCRIPTION:
Specific and validated instruments will be performed to women in their 8th week of postpartum period.

Those instruments are:

Edinburgh Postpartum Depression Scale (EPDS) Female genital self-image scale (FGSIS) Insomnia Severity Index (ISI) Breast-feeding efficacy scale short form (BSES-SF) Beck Depression Scale

ELIGIBILITY:
Inclusion Criteria:

* All women in the puerpera period (who gave consent)

Exclusion Criteria:

* None.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women who gave birth in Bartin State Hospital (the only one hospital in the city) after October 2018. for three months.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
Postpartum Depression | Change between the 4th, 8th and 12th weeks of postpartum period
  Postpartum Depression scores will be measured by Edinburgh Postpartum Scale (EDPS). The EDPS was developed to identify women who may have postpartum depression. Each answer is given a score of 0 to 3 . The maximum score is 30. The EPDS is a 10-item questionnaire. Women are asked to answer each question in terms of the past seven days. A score is calculated by adding the individual items as indicated A score of more than 10 suggests minor or major depression may be present.

SECONDARY OUTCOMES:
Genital self-image | At 4th, 8th and 12th week of postpartum period
  Genital Self-image scores will be measured by Female Genital Self Image Scale (FGSIS). FGSIS measures the genital self-image of the participants.
  The seven-item FGSIS assesses women's feelings and beliefs about their own genitals using a 4-point response scale (strongly agree, agree, disagree, strongly disagree).
  Respondents'scores on each item were summed for a total sum score ranging from 7 to 28, with higher scores indicating more positive genital self-image.
sleep disorders | At 4th, 8th and 12th week of postpartum period
  Sleep problems will be measured by Insomnia Severity Index (ISI). The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
breast-feeding | At 4th, 8th and 12th week of postpartum period
  Breast-feeding will be assessed by the Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF). It is a 14 item self-report instrument developed to measure a mother's perceived ability to breastfeed her infant. It has a five-point Likert scale for rating from 1 ("not at all confident") to 5 ("always confident"). Items ratings will be summed to produce a total score from 14 to 70, with higher scores indicating higher confidence. The means score points will be used as the cut-off point between high and low scorers.
socio-economic-demographical features | At 4th postpartum week
  Social, economic and demographic features will be assessed by a structured non-validated data gathering form

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yassa, MD, Principal Investigator — Bartin State Hospital
Locations (1):
- Bartin State Hospital, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lanes A, Kuk JL, Tamim H. Prevalence and characteristics of postpartum depression symptomatology among Canadian women: a cross-sectional study. BMC Public Health. 2011 May 11;11:302. doi: 10.1186/1471-2458-11-302. PMID 21569372